CLINICAL TRIAL: NCT05914012
Title: The Effects of Telerehabilitation Program Based on Otago Exercises on Balance, Frailty and Quality of Life in tOlder Adults: A Randomized-Controlled Study
Brief Title: Telerehabilitation Based on Otago Exercises for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Güzin Kara, PT. PhD. Assist. Prof., Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: E-60116787-020-136972
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Older Adults

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): 125 older adults aged 65 and over, who do not have any neurological, cognitive and communication problems that may affect the evaluations, and who volunteer to participate in the study and who are sedentary.
  Interventions: Other: Telerehabilitation based on Otago Exercise Program
- Control Group (No Intervention): 125 older adults not participating in any exercise program during the study, not having any neurological, cognitive and communication problems that may prevent completing the assessments.

INTERVENTIONS:
Other: Telerehabilitation based on Otago Exercise Program — It took a total of 21 sessions, 7 days a week for 3 weeks. The sessions lasted 30 minutes. It is recommended to do exercises with comfortable shoes at least 1 hour after a meal. Each of his exercises will be videotaped and numbered and delivered to the intervention group via social networks and the Internet or by memory. In each exercise session, the physiotherapist followed the exercise sessions through social networks and answered questions from the older adults.
  Arms: Intervention Group

SUMMARY:
This study is a single-blind, randomized controlled, prospective clinical trial. At least 62 older adults aged 65 and over were included in the study. Evaluations were made twice, before starting the study and after completion. Otago Exercise Program based on telerehabilitation was applied to the intervention group for a total of 21 sessions, 7 days a week for 3 weeks. The control group did not participate in any exercise program during the study period; however, it was reported that they could be included in the Otago Exercise Program at the end of the study.

DETAILED DESCRIPTION:
Sociodemographic data and information about falling were recorded. Edmonton Frail Scale, Modified Fall Efficiency Scale, Five-Dimensional European Quality of Life Scale-5D-3L, Timed Up and Go Test, Four-Step Balance Test and 30 sec Sit to StandTest were applied to all older adults. Evaluations were applied at the beginning and end of the study. A total of 21 sessions of Otago Exercise Program were applied to the intervention group, 30 minutes/session, 7 days/week for 3 weeks. A printed physical activity recommendation brochure prepared for the older adults by the Ministry of Health of the Republic of Turkey was distributed to both groups. The older adults in the control group did not participate in any exercise program during the study period.

ELIGIBILITY:
Inclusion Criteria for Intervention Group:

* Sedentary and sedentary older adults who do not have any neurological, cognitive, or communication problems that may affect assessments, and who volunteer to participate in the study.

Inclusion Criteria for Control Group:

* Not participating in any exercise program during the study, not having any neurological, cognitive and communication problems that may prevent completing the assessments.

Exclusion Criteria for Intervention Group:

* Participants who have communication problems, are younger than 65 years old, have any neurological diagnosis and have orthopedic, mental and communication problems that prevent evaluations, and do not consent to participate in the study.

Exclusion Criteria for Control Group:

* Those who do not meet the specified age criteria for the study, fail to complete the assessments, and continue the rehabilitation program.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — A web-based randomization program (https://www.randomizer.org/) will be used to randomize participants 1:1 to the intervention and control groups, stratified by gender.
Enrollment: 250 (Actual)
Dates: Start 2021-12-22 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
The Edmonton Frail Scale | 8 months
  The scale consists of nine areas of vulnerability, which are considered to be the determinants of vulnerability. Among these vulnerability areas, general health status and drug use are evaluated with two questions, and other areas with a single question. The scale consists of 11 items in total. Two areas of cognitive and functional performance are tested using performance-based items. Clock testing is used for cognitive status and timed up-and-go testing is used for functional performance. The test takes less than five minutes to administer. The minimum total score is zero and the maximum score is 17. An increase in the total score obtained from the scale indicates that the severity of vulnerability increases. fragility to scale; It consists of five levels: not fragile, sensitive, slightly fragile, moderately fragile, and severely fragile. The Turkish version of the scale was found to be valid and reliable.
The Modified Falls Efficacy Scale | 8 months
  The Modified Fall Efficiency Scale is an expanded version of the Fall Efficiency Scale, which includes items questioning confidence during 4 different outdoor activities. The scale evaluates the sense of security related to activities of daily living (such as dressing, bathing, crossing) on a ten-point visual analog scale. 10 items of the scale are related to indoor activities and 4 items are related to outdoor activities. Items in the scale are scored between 0 (not confident) and 10 (completely sure) to assess the participants' self-efficacy regarding falling. The scale score is calculated by dividing the sum of the scores per question by the number of questions. A high score means a high sense of safety and competence against falling. The Turkish validity and reliability study of the questionnaire was conducted.
The Five-Dimensional European Quality of Life Scale (EQ-5D-3L) | 8 months
  Consisting of five dimensions: movement, self-care, usual activities, pain/discomfort, and anxiety/depression, this scale was developed by the European Quality of Life Research Society (EuroQol) in 1990 to measure health-related quality of life. Each dimension of the scale is calculated over 3 points as no problem, some problem and major problem. In addition, individuals indicate their current health status by marking on a visual analog scale (0-100 points). The Turkish version was found to be valid and reliable.
The Timed Up and Go Test | 8 months
  The Timed Get Up and Go Test was developed in 1991 by Podsiadlo and Richardson. For the test, the individual is asked to get up from a standard chair, walk 3 meters, return and sit back in the chair. The duration begins with the individual getting up from the chair and ends with sitting down. The result is recorded in seconds.
The Four Step Balance Test | 8 months
  The test consists of four different tasks (feet together, semi-tandem, tandem, and standing on one leg) that become increasingly difficult in the standing position. After the patient regains his balance, the physiotherapist releases the support and the patient is asked to maintain the position. During this time, the time is kept and recorded in seconds. If the patient can hold the position for 10 seconds without moving his feet or needing support, the next position is passed.
The 30 sec Sit to Stand Test | 8 months
  The patient sits in a chair with a standard sitting height and backrest. They cross their hands on their chest. The patient is asked to sit and stand up from the chair as quickly as possible. The number of sitting and getting up is noted by keeping a 30-second timer with a stopwatch.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Kınıklı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen X, Zhao L, Liu Y, Zhou Z, Zhang H, Wei D, Chen J, Li Y, Ou J, Huang J, Yang X, Ma C. Otago exercise programme for physical function and mental health among older adults with cognitive frailty during COVID-19: A randomised controlled trial. J Clin Nurs. 2025 Dec;34(12):5130-5143. doi: 10.1111/jocn.15964. Epub 2021 Jul 21. PMID 34289524
- [Result] Binns E, Taylor D. The effect of the Otago Exercise Programme on strength and balance in community dwelling older women. New Zealand Journal of Physiotherapy. 2011;39(2).
- [Result] Agostini M, Moja L, Banzi R, Pistotti V, Tonin P, Venneri A, Turolla A. Telerehabilitation and recovery of motor function: a systematic review and meta-analysis. J Telemed Telecare. 2015 Jun;21(4):202-13. doi: 10.1177/1357633X15572201. Epub 2015 Feb 22. PMID 25712109